CLINICAL TRIAL: NCT02031991
Title: Phase 1, Double Blind, Randomized, Parallel-Group, Single-Dose, 3-Arm, Comparative Pharmacokinetic Study Of PF-06439535 And Bevacizumab Sourced From US And EU Administered To Healthy Male Volunteers
Brief Title: A Pharmacokinetic Study Comparing PF-06439535 And Bevacizumab In Healthy Male Volunteers (REFLECTIONS B739-01)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: B7391001; REFLECTIONS B739-01
Record Dates: First submitted 2014-01-07; First posted 2014-01-09 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2014-08

CONDITIONS: Healthy
Keywords: Bioequivalence; Biosimilarity; Similarity; PK; Phase 1; Bevacizumab; Healthy Volunteers; Single-Dose; Oncology
MeSH Terms: conditions — Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- A = PF-06439535 (Experimental): Intervention Description: Sterile vial 400mg, single-dose 5mg/kg administered as 90-minute infusion on day 1.
  Interventions: Biological: PF-06439535
- B = Bevacizumab-EU (Active Comparator): Intervention Description: Sterile vial 400mg, single-dose 5mg/kg administered as 90-minute infusion on day 1.
  Interventions: Biological: Avastin
- C = Bevacizumab-US (Active Comparator): Intervention Description: Sterile vial 400mg, single-dose 5mg/kg administered as 90-minute infusion on day 1.
  Interventions: Biological: Avastin

INTERVENTIONS:
Biological: PF-06439535 — Solution for intravenous infusion, single dose of 5mg/kg, administered as 90-minute infusion.
  Other Names: PF-06439535, a potential biosimilar to bevacizumab
  Arms: A = PF-06439535
Biological: Avastin — Solution for intravenous infusion, single dose of 5mg/kg, administered as 90-minute infusion.
  Other Names: Bevacizumab (European Union)
  Arms: B = Bevacizumab-EU
Biological: Avastin — Solution for intravenous infusion, single dose of 5mg/kg, administered as 90-minute infusion.
  Other Names: Bevacizumab (United States)
  Arms: C = Bevacizumab-US

SUMMARY:
This study is to prove that the handling (also referred to as pharmacokinetics) of the following drugs PF-06439535, Avastin® (bevacizumab) that is licensed for use in the United States (bevacizumab-US) and Avastin® (bevacizumab) obtained from Europe (bevacizumab-EU) is similar in healthy male volunteers after receiving a single intravenous dose of either drugs.

During the course of the study, the similarity in pharmacokinetics will be assessed by sampling the levels of drug in the blood, and by comparing these levels among the different administration arms of PF-06439535, bevacizumab-US and bevacizumab-EU. Safety, tolerability, and immunologic response to the administered drugs will also be evaluated throughout.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects 21-55 years old
* Subjects who have previously been exposed to a biologic agent (other than a VEGF [Vascular Endothelial Growth Factor Receptor] inhibitor) may enroll provided that at least 3 months have passed since the last administration of that drug
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50kg (110lbs)

Exclusion Criteria:

* Evidence or history of a clinically significant disease or clinical finding at Screening
* Previous treatment with an anti-VEGF antibody, or any other antibody or protein targeting the VEGF receptor.

Ages: 21 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2014-01; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | Day 1 - Day 71
Area Under the Curve from Time Zero to end of dosing interval (AUCtau) | Day 1 - Day 71
Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - 8)] | Day 1 - Day 71
  AUC (0 - 8)= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - 8). It is obtained from AUC (0 - t) plus AUC (t - 8).

SECONDARY OUTCOMES:
Systemic Clearance (CL) | Day 1 - Day 71
Terminal Disposition Half-Life (t1/2) | Day 1 - Day 71
Volume of Distribution at Steady State (Vss) | Day 1 - Day 71
Incidence of anti-bevacizumab antibodies (ADA), including neutralizing antibodies (Nab) | Day 1 - Day 71 or LSLV, whichever occurs later

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, South Miami, Florida, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7391001&StudyName=A%20Pharmacokinetic%20Study%20Comparing%20PF-06439535%20And%20Bevacizumab%20In%20Healthy%20Male%20Volunteers%20%28REFLECTIONS%20B739-01%29